CLINICAL TRIAL: NCT01722162
Title: Phase II Study of Levocetirizine in Combination With Capecitabine + Bevacizumab to Overcome Resistance to Anti-angiogenic Therapy in Patients With Refractory Colorectal Cancer
Brief Title: Levocetirizine + Capecitabine + Bevacizumab for Patients With Refractory Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201303043
Record Dates: First submitted 2012-10-29; First posted 2012-11-06 (Estimated); Results first posted 2017-02-13 (Actual); Last update posted 2017-04-20 (Actual); Status verified 2017-03

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Capecitabine; levocetirizine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A: (start levocetirizine after bevacizumab/capecitabine) (Experimental): Bevacizumab IV 5 mg/kg on Days 1 each 2-week cycle.
  Capecitabine PO 850 mg/m2 twice a day on Days 1-7 of each 2 week cycle.
  Levocetirizine PO 5 mg daily before bed starting on Day 8 of Cycle 1. 5 mg daily before bed Days 1-4 of each cycle starting with cycle 2.
  Interventions: Drug: Bevacizumab; Drug: Capecitabine; Drug: Levocetirizine
- Arm B: (start levocetirizine before bevacizumab/capecitabine) (Experimental): Bevacizumab IV 5 mg/kg on Days 1 each 2-week cycle.
  Capecitabine PO 850 mg/m2 twice a day on Days 1-7 of each 2 week cycle.
  Levocetirizine PO 5 mg daily starting 7 days prior to initiation of bevacizumab and capecitabine therapy. 5 mg daily Days 1-14 starting with cycle 2.
  Interventions: Drug: Bevacizumab; Drug: Capecitabine; Drug: Levocetirizine

INTERVENTIONS:
Drug: Bevacizumab
  Other Names: Avastin®
Drug: Capecitabine
  Other Names: Xeloda®
Drug: Levocetirizine
  Other Names: Xyzal

SUMMARY:
This randomized phase II trial studies how giving a drug called levocetirizine to patients with colorectal cancer affects their tumor response to capecitabine and bevacizumab. Capecitabine is a chemotherapy drug that blocks tumor growth by disrupting DNA and RNA synthesis and repair (cell division and survival). Bevacizumab is a monoclonal antibody that blocks the ability of tumors to grow and spread by inhibiting the growth of blood vessels that feed them. Patients with colorectal cancer can develop a resistance to the effects of bevacizumab. Levocetirizine may decrease tumor resistance to bevacizumab. Giving bevacizumab, capecitabine, and levocetirizine dihydrochloride together may be an effective treatment for refractory colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have histologically or cytologically confirmed refractory colorectal cancer (CRC).
* Patient must have measurable disease defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥10 mm with CT scan, as ≥20 mm by chest x-ray, or ≥10 mm with calipers by clinical exam.
* Patient must have documented progressive disease within 3 months of his/her most recent cycle of chemotherapy.
* Patient must be refractory to or intolerant of prior therapy with a fluoropyrimidine, oxaliplatin, irinotecan, and/or anti-angiogenic therapy. Patients with K-RAS wild type tumors must have received an epidermal growth factor receptor (EGFR) inhibitor such as cetuximab or panitumumab.
* Patient must be ≥ 18 years of age.
* Patient must have an ECOG performance status ≤ 2
* Patient must have normal bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1,500/mcl
  * Platelets ≥ 100,000/mcl
  * Total bilirubin ≤ 2.0 x IULN
  * AST(SGOT)/ALT(SGPT) ≤ 3.0 x IULN
  * Patients must have adequate renal function prior to chemotherapy defined as serum creatinine ≤ 2.0 mg/dl OR Creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with creatinine levels above 2.0
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Patient must be able to understand and willing to sign an IRB approved written informed consent document.

Exclusion Criteria:

* Patient must not have a history of other malignancy ≤ 3 years previous with the exception of basal cell or squamous cell carcinoma of the skin which were treated with local resection only or carcinoma in situ of the cervix.
* Patient must not be receiving any other investigational agents.
* Patient must not have known active brain metastases. Patients with previously treated brain metastases are eligible. Patients with known brain active metastases must be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Patient must not have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to levocetirizine, capecitabine, bevacizumab, or other agents used in the study.
* Patient must not have known dihydropyrimidine dehydrogenase (DPD) deficiency or severe renal impairment (creatinine clearance below 30 mL/min by Cockcroft and Gault formula) as this would prelude use of capecitabine.
* Patient must not have known proteinuria ≥ 500mg/24 hours.
* Patient must not have an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patient must not be pregnant and/or breastfeeding. Patient must have a negative urine pregnancy test within seven days of study entry.
* Patient must not be known to be HIV-positive on combination antiretroviral because of the potential for pharmacokinetic interactions with levocetirizine, capecitabine, and bevacizumab. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2013-04; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manik A Amin, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to patient enrollment on 04/26/2013 and closed to patient enrollment on 07/15/2015.
Period: Overall Study
Arm/Group | Arm A: (Start Levocetirizine After Bevacizumab/Capecitabine) | Arm B: (Start Levocetirizine Before Bevacizumab/Capecitabine)
Started | 23 | 24
Completed | 18 | 18
Not Completed | 5 | 6
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Found ineligible | 1 | 0
Not completed — Unrelated to study adverse event | 2 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Insurance denial post enrollment | 0 | 1
Not completed — Noncompliance | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: (Start Levocetirizine After Bevacizumab/Capecitabine) | Arm B: (Start Levocetirizine Before Bevacizumab/Capecitabine) | Total
Number analyzed (Participants) | 23 | 24 | 47
Age, Continuous [Median (Full Range); unit: years] | 62 [39 to 80] | 57.5 [36 to 76] | 60 [36 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 14 | 15 | 29
Region of Enrollment [Number; unit: participants]
  United States | 23 | 24 | 47

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (Arm A)
Description: * Time from start of treatment to the time of progression or death, whichever occurs first
  * Progressive disease (target lesions): at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
  * Progressive disease (non-target lesions): appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Time Frame: Until progressive disease (PD) (estimated to be 92 days)
Measure: Number (95% Confidence Interval); unit: proportion of patients with PFS
Arm/Group | Arm A: (Start Levocetirizine After Bevacizumab/Capecitabine)
Number analyzed (Participants) | 18
proportion of patients with PFS
  PFS Days = 29 | 0.946 [0.848 to 1.00]
  PFS Days = 36 | 0.892 [0.761 to 1.00]
  PFS Days = 43 | 0.739 [0.567 to 0.964]
  PFS Days = 46 | 0.685 [0.505 to 0.929]
  PFS Days = 50 | 0.630 [0.446 to 0.890]
  PFS Days = 92 | 0.575 [0.390 to 0.849]

2. Secondary Outcome: Incidence and Severity of Adverse Events as Measured by Number of Participants Who Experience Grade 3 and Higher Adverse Events
Description: NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Time Frame: Up to 6 months
Population: Arm A: 4 patients not evaluable for outcome measure (2 had unrelated adverse events after enrollment but prior to treatment, 1 withdrew consent after enrollment but prior to treatment, & 1 was found ineligible after enrollment but prior to treatment). Arm B: 1 patient not evaluable because of noncompliance after enrollment but before treatment
Measure: Number; unit: participants
Arm/Group | Arm A: (Start Levocetirizine After Bevacizumab/Capecitabine) | Arm B: (Start Levocetirizine Before Bevacizumab/Capecitabine)
Number analyzed (Participants) | 19 | 23
participants
  Small intestinal obstruction | 1 | 0
  Fatigue | 1 | 1
  Urinary tract infection | 1 | 0
  Blood bilirubin increased | 2 | 0
  Peripheral motor neuropathy | 1 | 0
  Peripheral sensory neuropathy | 1 | 0
  Dyspnea | 1 | 2
  Hypertension | 1 | 2
  Thromboembolic event | 1 | 0
  Anemia | 0 | 1
  Heart failure | 0 | 1
  Colonic fistula | 0 | 1
  Colonic perforation | 0 | 1
  Gram-negative bacilli infection | 0 | 1
  Clostridium bloodstream infection | 0 | 1
  Alanine aminotransferase increased | 0 | 1
  Anorexia | 0 | 1
  Bone pain | 0 | 1
  Generalized muscle weakness | 0 | 1
  Muscle weakness lower limbs | 0 | 1
  Urinary retention | 0 | 1
  Respiratory failure | 0 | 1

3. Primary Outcome: Progression Free Survival (Arm B)
Description: as for outcome 1
Time Frame: Until progressive disease (PD) (up to 60 days)
Measure: Number (95% Confidence Interval); unit: proportion of patients with PFS
Arm/Group | Arm A: (Start Levocetirizine After Bevacizumab/Capecitabine)
Number analyzed (Participants) | 18
proportion of patients with PFS
  PFS Days = 29 | 0.946 [0.848 to 1.00]
  PFS Days = 33 | 0.892 [0.761 to 1.00]
  PFS Days = 44 | 0.838 [0.686 to 1.00]
  PFS Days = 50 | 0.686 [0.507 to 0.928]
  PFS Days = 54 | 0.631 [0.448 to 0.890]
  PFS Days = 60 | 0.576 [0.391 to 0.849]

ADVERSE EVENTS:
Description: Arm A: 4 patients not evaluable for serious adverse event and adverse event collection (2 had unrelated adverse events after enrollment but prior to treatment, 1 withdrew consent after enrollment but prior to treatment, & 1 was found ineligible after enrollment but prior to treatment). Arm B: 1 patient not evaluable for serious adverse event and adverse event collection because of noncompliance after enrollment but before treatment
Arm/Group | Arm A: (Start Levocetirizine After Bevacizumab/Capecitabine) | Arm B: (Start Levocetirizine Before Bevacizumab/Capecitabine)
Serious Adverse Events (participants affected / at risk) | 5/19 | 6/23
Other Adverse Events (participants affected / at risk) | 19/19 | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: (Start Levocetirizine After Bevacizumab/Capecitabine) (N=19) | Arm B: (Start Levocetirizine Before Bevacizumab/Capecitabine) (N=23)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Colonic fistula (Gastrointestinal disorders) | 0 | 1
Illeal hemorrhage (Gastrointestinal disorders) | 1 | 0
Small bowel obstruction (Gastrointestinal disorders) | 1 | 0
Death due to disease progression (General disorders) | 2 | 2
Generalized weakness (General disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute renal failure (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: (Start Levocetirizine After Bevacizumab/Capecitabine) (N=19) | Arm B: (Start Levocetirizine Before Bevacizumab/Capecitabine) (N=23)
Anemia (Blood and lymphatic system disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Watering eyes (Eye disorders) | 0 | 1
Abdominal cramps (Gastrointestinal disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 3
Bleeding at stroma site (Gastrointestinal disorders) | 0 | 1
Bloating (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Colonic perforation (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 3 | 8
Dehydration (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 9 | 9
Dry mouth (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 4
Flatulence (Gastrointestinal disorders) | 0 | 1
Hemmorrhoids (Gastrointestinal disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 4 | 5
Nausea (Gastrointestinal disorders) | 4 | 11
Oral hemorrhage (Gastrointestinal disorders) | 3 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1
Stomach pain (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 5 | 23
Chills (General disorders) | 3 | 2
Edema - limbs (General disorders) | 3 | 3
Fatigue (General disorders) | 11 | 11
Fever (General disorders) | 2 | 2
Flu-like symptoms (General disorders) | 1 | 0
Gait disturbance (General disorders) | 1 | 0
Localized edema (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Pain (General disorders) | 5 | 1
Sweating (General disorders) | 1 | 0
Bronchial infection (Infections and infestations) | 1 | 0
Clostridium bloodstream infection (Infections and infestations) | 0 | 1
Food poisoning "stomach flu" (Infections and infestations) | 1 | 0
Gastroenteritis (Gastrointestinal disorders) | 1 | 0
Gram-negative bacilli infection (Infections and infestations) | 0 | 1
Lip infection (Infections and infestations) | 0 | 1
Otitis externa (Infections and infestations) | 1 | 0
Right groin infection (Infections and infestations) | 0 | 1
Shingles (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 1 | 1
Upper respiratory infection (Infections and infestations) | 3 | 2
Urinary tract infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Alkaline phosphatase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 2
Blood bilirubin increased (Investigations) | 3 | 1
Hypoalbuminemia (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 2 | 1
Weight loss (Investigations) | 2 | 0
White blood cell decreased (Investigations) | 2 | 0
Anorexia (Metabolism and nutrition disorders) | 6 | 7
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cramping in hands and feet (Musculoskeletal and connective tissue disorders) | 1 | 0
Foot pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle cramps (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness lower limbs (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 3 | 3
Dysgeusia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 7 | 3
Neuralgia (Nervous system disorders) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 5 | 3
Presyncope (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 2
Confusion (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 2
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Dry nasal passages (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Trachypneic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Brittle nails (Skin and subcutaneous tissue disorders) | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 3
Facial rash (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar-Planter erythrodysethsia (Skin and subcutaneous tissue disorders) | 3 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 2
Skin pain (Skin and subcutaneous tissue disorders) | 1 | 0
Sores on head (Skin and subcutaneous tissue disorders) | 1 | 0
Cataract surgery (Surgical and medical procedures) | 0 | 1
Hot flashes (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 2 | 2
Thromboembolic event (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes